CLINICAL TRIAL: NCT05535491
Title: The Effection Pain and Anxiety of a Breathing Exercise Applied Following Laparoscopic Cholecystectomy: A Randomized Controlled Study
Brief Title: The Effection Pain and Anxiety of a Breathing Exercise Applied Following Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Aylin Aydin Sayilan, Associate Professor, Kırklareli University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P0115R00
Record Dates: First submitted 2022-09-02; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1 (Experimental): BREATHING EXERCISE GROUP
  Interventions: Other: Educational and Research Hospital
- GROUP 2 (No Intervention): CONTROL GROUP

INTERVENTIONS:
Other: Educational and Research Hospital — breathing exercise
  Arms: GROUP 1

SUMMARY:
One important part of individual nursing care is that that nurses teach and apply breathing exercises, which are vital and increase the patient's quality of life, in the light of their current knowledge and skills. The purpose of this study was therefore to determine the effect of postoperative breathing exercises on pain and anxiety in patients hospitalized in the general surgery clinic and who had undergone laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Introduction: Several methods are employed for overcoming pain and anxiety that are frequently experienced in the postoperative period. This study was planned to determine the effect of a breathing exercise on patient pain and anxiety after laparoscopic cholecystectomy.

Methods: The sample determined using power analysis in this randomized, controlled, semi-experimental research performed in two hospitals in the west of Turkey between January and November 2019 consisted of 74 individuals (37 experimental and 37 controls). An information form involving descriptive characteristics, a visual analogue scale (VAS), and the State-Trait Anxiety Inventory (STAI I/II) were used for data collection. Descriptive statistical methods and parametric tests were employed in the data analysis.

ELIGIBILITY:
Inclusion Criteria

* Hospitalized in the general surgery clinics,
* with histories of laparoscopic cholecystectomy,
* consenting to take part.

Exclusion Criteria:

- Have a psychiatric disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Postoperative anxiety scores would be lower in the experimental group than in the control group. | six months
  Postoperative anxiety scores
Postoperative pain score would be lower in the experimental group than in the control group. | six months
  Postoperative pain score

CONTACTS AND LOCATIONS:
Overall Officials: Aylin AYDIN SAYILAN, PhD, Study Chair — Kırklareli University
Locations (1):
- Lüleburgaz Devlet Hastanesi, Kırklareli, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koras K, Karabulut N. The Effect of Foot Massage on Postoperative Pain and Anxiety Levels in Laparoscopic Cholecystectomy Surgery: A Randomized Controlled Experimental Study. J Perianesth Nurs. 2019 Jun;34(3):551-558. doi: 10.1016/j.jopan.2018.07.006. Epub 2018 Nov 20. PMID 30470466
- [Background] Saritas S, Genc H, Okutan S, Inci R, Ozdemir A, Kizilkaya G. The Effect of Comedy Films on Postoperative Pain and Anxiety in Surgical Oncology Patients. Complement Med Res. 2019;26(4):231-239. doi: 10.1159/000497234. Epub 2019 Mar 27. PMID 30921794
- [Background] Sao CH, Chan-Tiopianco M, Chung KC, Chen YJ, Horng HC, Lee WL, Wang PH. Pain after laparoscopic surgery: Focus on shoulder-tip pain after gynecological laparoscopic surgery. J Chin Med Assoc. 2019 Nov;82(11):819-826. doi: 10.1097/JCMA.0000000000000190. PMID 31517775
- [Background] Santivanez-Acosta R, Tapia-Lopez ELN, Santero M. Music Therapy in Pain and Anxiety Management during Labor: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2020 Oct 10;56(10):526. doi: 10.3390/medicina56100526. PMID 33050409
- [Background] Ju W, Ren L, Chen J, Du Y. Efficacy of relaxation therapy as an effective nursing intervention for post-operative pain relief in patients undergoing abdominal surgery: A systematic review and meta-analysis. Exp Ther Med. 2019 Oct;18(4):2909-2916. doi: 10.3892/etm.2019.7915. Epub 2019 Aug 19. PMID 31555379